CLINICAL TRIAL: NCT00186368
Title: Microarray Analysis of Gene Expression in Prostate Tissues (Translating Prostate Cancer Gene Expression Sub-types)
Brief Title: Microarray Analysis of Gene Expression in Prostate Tissues
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Wisconsin, Madison (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James D Brooks, Professor Clinical (Primary) Uro-Oncology, Stanford University
Other Study IDs: PROS0009; PROS0009 (Other: Stanford University); 13873 (Other: Stanford IRB); 1U01CA196387 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Gene expression; tumor markers; microarray analysis
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate gene expression profiles and biologic features of prostate tissue and how they relate to prostate cancer development and growth.

ELIGIBILITY:
Inclusion Criteria:

- Patient scheduled to undergo either a biopsy or surgery for a prostate condition.

Exclusion Criteria:

- Patients without a prostate condition

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Per the original application in 1999: After obtaining informed consent (via the Tissue Bank consent), Protocol # 13873 (Continuing Review) PROTOCOL Print Date: September 22, 2010 PD: James Duane Brooks APPLICATION FORM Page 11 of 22 Review Type: Expedited Human Subjects Research Medical Stanford University Title: Microarray Analysis of Gene Expression in Prostatic Tissues (SQL 76528) Approval Period: 07/31/2010 - 06/30/2011 specimens will be collected from the Stanford University Department of Pathology (Tissue Bank) for patients treated at Stanford. Patients will be followed up via chart or tumor registries. Data will be used strictly for research purposes. Gene expression arrays are done in Dr. Brook's laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 867 (Actual)
Dates: Start 1999-04-06 (Actual); Primary Completion 2009-04-21 (Actual); Study Completion 2009-04-21 (Actual)

PRIMARY OUTCOMES:
Correlate genotype with pathologic phenotype and clinical outcome. | one time
  The Tissue Bank will store all "Tissue Bank" consents. The patients will be given a unique identifier by the tissue bank. However, patients will need to be identified to link to clinical data and possible followup (if they have consented) via chart or tumor registries.

CONTACTS AND LOCATIONS:
Overall Officials: James Brooks, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Cancer Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No